CLINICAL TRIAL: NCT03707223
Title: Evaluating the Effectiveness of "The Interfaces Program" to Promote Person's Components, Performance and Improving the Work Environment of People With Disabilities
Brief Title: Effectiveness of Interfaces Program to Promote Work Ability of People With Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Laszlo Tauber Family Foundation (Unknown)
Responsible Party: Principal Investigator, Navah Ratzon, Professor, Occupational Therapist, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Maya Huber; Principal Investigator (Prof) (Other: TelAvivU); Principal Investigator (Other: TelAvivU)
Record Dates: First submitted 2017-04-29; First posted 2018-10-16 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Disabilities Mental; Disabilities Physical
Keywords: career development, people with disabilities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental (Experimental): The "interfaces Program"
  Interventions: Behavioral: The Interfaces Program
- control group (Active Comparator): supported employment using the individual placement and support (IPS) model
  Interventions: Behavioral: IPS

INTERVENTIONS:
Behavioral: The Interfaces Program — career development program
  Arms: experimental
Behavioral: IPS — supported employment using the individual placement and support (IPS) model
  Arms: control group

SUMMARY:
the objectives of the study is to Evaluate the effectiveness of "The Interfaces Program" to promote person's components, performance and improving the work environment of people with disabilities.

DETAILED DESCRIPTION:
People with disabilities experience many barriers in trying to integrate into the competitive market. The barriers may be result of the unique characteristics of the individual (characteristics of the disability, occupational history, work self-efficacy, etc.), the characteristics of the occupation and occupational performance (characteristics of the job and the job demands) and environmental barriers (accessibility, discrimination, stigma and lack of opportunities, etc.). The main response to the integration problems of people with disabilities in the world of work is supported employment service. Supported employment focuses primarily on placement of the individual and do not relate to barriers relating to the individual's ability to develop a career.

The present study examines the effectiveness of a new intervention program "The interfaces program " aiming to promote career development process among people with disabilities working in the competitive market. The program presents an integration of the Person-Environment-Occupation-Performance (PEOP) model and lead career development theories. The ultimate goal of this study is to examine the effectiveness of the "interfaces program" by examining its impact on the promotion of objective and subjective measures among people with disabilities who work and receive supported employment services.

ELIGIBILITY:
Inclusion Criteria:

* psychiatric or physical disability
* 12 years of educations minimum
* at least 26 score on the Montreal cognitive assessment ( MOCA)
* working at least 3 month in the open market

Exclusion Criteria:

* autistic spectrum disorder (ASD)
* Developmental Cognitive Disability
* alcohol or drags comorbidities

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-09; Primary Completion 2018-08 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
proactive behavior Questionnaire (developed for this study) | A change in proactive behavior measure will appear after 9 sessions over 3 month (4 first meeting will be done once a week, and 5 meetings once in two weeks) of intervention, and after 3 month form the end of the intervention
  proactive behavior during the last week
Adult subjective assessment of participation (ASAP) | A change in subjective experience of participation measure will appear after 9 sessions over 3 month (4 first meeting will be done once a week, and 5 meetings once in two weeks) of intervention, and after 3 month form the end of the intervention
  subjective experience of participation in meaningful occupations
Work Behavior Inventory (WBI) | A change in work behavior measure will appear after 9 sessions over 3 month (4 first meeting will be done once a week, and 5 meetings once in two weeks) of intervention, and after 3 month form the end of the intervention
  employer assessment of work behavior and work performance
work self efficacy Questionnaire (WSS-37) | A change in work self efficacy measure will appear after 9 sessions over 3 month (4 first meeting will be done once a week, and 5 meetings once in two weeks) of intervention, and after 3 month form the end of the intervention
  subjective report of work self efficacy
health perception sf 12 Questionnaire Health Perception | A change in health perception measure will appear after 9 sessions over 3 month (4 first meeting will be done once a week, and 5 meetings once in two weeks) of intervention, and after 3 month form the end of the intervention
  subjective report of health perception
career self management - subjective self management perception Questionnaire - developed for this study | A change in career self management measure will appear after 9 sessions over 3 month (4 first meeting will be done once a week, and 5 meetings once in two weeks) of intervention, and after 3 month form the end of the intervention
  subjective report of career self management
perception of environmental work barriers - subjective work barriers perception Questionnaire - developed for this study | A change in perception of environmental barriers will appear after 9 sessions over 3 month (4 first meeting will be done once a week, and 5 meetings once in two weeks) of intervention, and after 3 month form the end of the intervention
  subjective perception of environmental work barriers

CONTACTS AND LOCATIONS:
Overall Officials: navah ratzon, prof, Principal Investigator — Tel Aviv University; Rachel Gali cinamonp, prof, Principal Investigator — Tel Aviv University
Locations (1):
- Maya Huber, Tel Aviv, Isarel, Israel

IPD SHARING:
Plan to Share IPD: No